CLINICAL TRIAL: NCT03153306
Title: Importance of the Infusion Rate for the Plasma Expanding Effect of 5% Albumin in the Septic Patient
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hainan People's Hospital (Other)
Collaborators: Southern Medical University, China (Other)
Responsible Party: Principal Investigator, rui li, Attending Doctor, critical care medicine department, Hainan People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HannanPH
Record Dates: First submitted 2016-05-17; First posted 2017-05-15 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Sepsis
Keywords: Albumin
MeSH Terms: conditions — Sepsis | interventions — Albumins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- the "bolus" group (Experimental): 10ml/kg of the natural colloid 5% albumin was given at 1 hrs.
  Interventions: Drug: albumin
- the"continuous" group (Experimental): 10ml/kg of the natural colloid 5% albumin was given over 6 hrs
  Interventions: Drug: albumin

INTERVENTIONS:
Drug: albumin — Two groups were formed at random for each fluid. In one group, 10ml/kg of 5% albumin was given over 1 hour (the "bolus" group), and in the other group, the same volume was given over 6 hrs (the"continuous" group)
  Other Names: human albumin(Austria)

SUMMARY:
Correction of hypovolemia is an important therapeutic measure，Even though there is no consensus regarding infusion rates, a plasma volume (PV) expander is often given at a fast rate to treat a suspected hypovolemia without delay which can be associated with aggravation of adverse interstitial accumulation of macromolecules and fluid, especially in inflammatory conditions such as sepsis.the smallest possible volumes for PV resuscitation to maintain normovolemia should be used to reduce the risk of simultaneous interstitial fluid accumulation. The investigators tested the hypothesis that a slow infusion rate of a PV expander results in better plasma expansion than a fast infusion rate to patients with severe sepsis or septic shock.

ELIGIBILITY:
Inclusion Criteria:

* admitted to the ICU patients with severe sepsis or septic shock (diagnosis according to the 2012 surviving sepsis campaign guidelines)
* there is low blood pressure (SBP < 90 or mean arterial pressure(MAP) < 65 or the systolic blood pressure is decreased 40 mmHg more than the basic level) or lactic acid or greater for 4 mmol/l
* the informed consent

Exclusion Criteria:

* less than 18 years of age
* more than 80 years old
* pregnant women
* albumin allergies
* the dying patients expected lifetime no more than 24 hours)
* patient with myocardial infarction, heart failure
* liver failure
* refused to sign the informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-06 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Extravascular lung water (EVLW) before and after fluid resuscitation | 6 hour
  Extravascular lung water （EVLW）is measured by Pulse index continous cardiac output (PICCO) before and after fluid resuscitation in each group

CONTACTS AND LOCATIONS:
Locations (1):
- Hainan Provincial People'S Hospital, Haikou, Hainan, China

IPD SHARING:
Plan to Share IPD: Yes